CLINICAL TRIAL: NCT07061769
Title: Evaluating the Safety and Effectiveness of a Low Intensity Cranial PEMF Device in Improving Chemotherapy Induced Peripheral Neuropathy Symptoms
Brief Title: Helping Cancer Patients Manage Neuropathy Symptoms From Chemotherapy With a Low-Intensity, Low-Risk Cranial PEMF Device
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: FluxWear, INC (Industry)
Collaborators: Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1391997
Record Dates: First submitted 2025-06-23; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Chemotherapy Induced Peripheral Neuropathy; Chemotherapy Induced Peripheral Neuropathy (CIPN); Chemotherapy Induced Pain Neuropathy; Chemotherapy Induced Neuropathic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment Device (Experimental)
  Interventions: Device: SHIFT
- Sham Device (Sham Comparator)
  Interventions: Device: SHIFT

INTERVENTIONS:
Device: SHIFT — SHIFT is a low intensity PEMF cranial device. It has been designated as a Non-Significant Risk device by the FDA.

SUMMARY:
The goal of this clinical trial is to examine a low-intensity, low-risk cranial PEMF device and its effectiveness with helping cancer patients manage neuropathy symptoms from chemotherapy. Eligible patients are individuals who have been diagnosed with chemotherapy-induced peripheral neuropathy or are experiencing pain due to chemotherapy and are eighteen to sixty. The main questions the study aims to answer are:

To examine whether the application of low intensity, low frequency PEMF (by the System for Heterogeneous Integrated magnetic Field Transmission (SHIFT)) results in a significant decrease in neuropathic pain intensity.

To examine if SHIFT results in a decrease of pain related interference and associated symptoms of CIPN.

Researchers will compare an active, treatment arm to a placebo, SHAM arm. Participants will be required to use the device once daily, fill out daily, weekly, and monthly surveys. They will have to do one blood draw at the beginning of the study and one at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Able to use smart phone and willing to receive text messages/emails
* Has CIPN disorder/neuropathic pain related to chemotherapy
* Able and willing to follow instructions
* Not participated in any other clinical study within the past two months that may influence the results of this study

Exclusion Criteria:

* History of seizures
* Hydrocephalic
* Had a change in medical therapy related to the treatment of neuropathy or chronic pain in the last fourteen days
* Received repetitive transcranial magnetic stimulation (rTMS) in the last 60 days
* Implanted device or metal in the brain
* History of brain bleed in the last six months
* History of suicidal behavior, bipolar disorder, schizophrenia
* Active radiation over the scalp
* Brain metastases
* Currently participates in other neuropathic pain studies
* Has any other medical condition that would prevent them from participating, including scalp wounds, hyperhidrosis, sensitive scalp, rash
* Pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Decrease in Neuropathic Pain Intensity | 12 weeks
  Measured through scores in the Neuropathy Pain Scale. The Neuropathy Pain Scale uses a range a 0 to 10, with 0 being no pain/sensation and 10 being the most intense pain/sensation imaginable.
Decrease in Numeric Pain Rating. | 12 weeks
  Measured through Numeric Pain Rating surveys. The numeric pain rating scale uses a range of 0 to 10, with 0 being no pain and 10 being the worst pain possible.
Improvement in Neuropathic Pain Symptoms | 12 weeks
  Measured in weekly scores in the Neuropathic Pain Symptom Inventory. The inventory uses a scale of 1 to 10, with 1 being the no symptom and 10 being the worst symptom imaginable.

SECONDARY OUTCOMES:
Decrease of pain-related interference | 12 weeks
  Examine if SHIFT results in a decrease of pain related interferences on a weekly basis. The PEG scale assesses how much pain interferes with weekly abilities on a scale of 0 to 10, with 0 being no interference/pain and ten being complete interference/worst pain imaginable.
Decrease of pain-related stress | 12 weeks
  Examine if SHIFT results in a decrease of perceived stress related to pain on a weekly basis, using the perceived stress scale. The PSS examines how well patients have been able to sleep on a scale of 0 to 4 (0 being never and 4 being very often).
Decrease of pain-related anxiety | 12 weeks
  Examine if SHIFT results in a decrease of anxiety related to pain as measured by the GAD-7. The GAD 7 uses a scale of 0 (not at all) to 3 (nearly every day) to measure how often a patient feels anxiety.
Decrease of pain-related inflammatory markers | 12 weeks
  Examine if SHIFT results in a decrease of inflammatory markers in the blood, specifically a decrease in the presence of IL-6.

CONTACTS AND LOCATIONS:
Locations (1):
- Hoag Spine Institute, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: Undecided